CLINICAL TRIAL: NCT04106180
Title: An Open-label, Multicenter, Phase II Single Arm Trial of SBRT in Combination With Sintilimab and GM-CSF for the Treatment of Advanced NSCLC
Brief Title: SBRT in Combination With Sintilimab and GM-CSF for the Treatment of Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sword
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sintilimab; Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT + sintilimab + GM-CSF (Experimental)
  Interventions: Drug: GM-CSF; Drug: Sintilimab; Radiation: SBRT

INTERVENTIONS:
Drug: GM-CSF — Patients will receive GM-CSF 125μg/m2 daily for 14 consecutive days after completing SBRT treatment.
Drug: Sintilimab — Patients will receive Sintilimab 200 mg every 3 weeks up to 2 years after completing SBRT treatment.
Radiation: SBRT — Patients will receive SBRT for one previously unirradiated primary or metastatic lesion (size: 1-5cm). 24 Gy in 3 fractions (8Gy/Fx) administered once-daily for 3 consecutive days.
  Other Names: Stereotactic body radiation therapy

SUMMARY:
This study is an open-label, multicenter, phase II single arm trial to evaluate the efficacy and safety of SBRT in combination with sintilimab and GM-CSF for the treatment of patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years.
* ECOG PS 0-1.
* Pathologically confirmed stage IV NSCLC.
* Negative for driver genes including EGFR，ALK，and ROS-1.
* Patients with disease progression after first-line platinum-based therapy without anti-PD-1 or PD-L1 treatment.
* Patients with at least one lesion (size 1-5cm) eligible for SBRT (24Gy/3Fx) and simultaneously at least one measurable lesion (in addition to the lesion treated with SBRT) as defined by RECIST1.1.
* Patients with brain metastasis are eligible if they are asymptomatic, neurologically stable, and off corticosteroids.
* Life expectancy of more than 3 months.
* Patients with no indications for palliative radiotherapy in the opinion of the investigator.
* Patients with a prior history of surgery are eligible if they have recovered adequately from the toxicity and/or complications of surgery.
* Signed informed consent for the use of fresh tumor biopsies before and during the treatment.
* Women of childbearing age and men must agree to use effective contraception during the trial.
* Adequate organ function within 1 week prior to the enrollment：

  1. Adequate bone marrow function: hemoglobin ≥80g/L, white blood cell (WBC) count ≥ 4.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, and platelet count ≥ 100 * 10 ^ 9/L;
  2. Adequate hepatic function: total bilirubin < 1.5 x upper limit of normal (ULN). Note: If total bilirubin is > 1.5 x ULN, direct bilirubin must ≤ ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 ULN;
  3. Adequate renal function: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min;
* Ability to understand and willingness to provide the informed consent.

Exclusion Criteria:

* Prior exposure to immunomodulatory agent,including but limited to anti-PD-1 or anti-PD-L1 antibodies.
* Severe autoimmune disease: inflammatory bowel disease (including Crohn's disease and ulcerative colitis) 、rheumatoid arthritis、scleroderma、systemic lupus erythematosus 、Wegener's granulomatosis and related vasculitides.
* Patients receiving non-platinum-based chemotherapy as first-line treatment
* Mixed small cell with non-small cell lung cancer histology.
* Pregnant or lactating women.
* Symptomatic interstitial lung disease or active infectious/non-infectious pneumonitis.
* History of any other malignancy.
* Patients in whom palliative radiotherapy is indicated in the opinion of the investigator.
* Active infection, congestive heart failure, myocardial infarction within the 6 months prior to enrollment, unstable angina pectoris or cardiac arrhythmia.
* Prior allergic reaction or contraindications to sintilimab and GM-CSF.
* Patients who have received tumor vaccine; or administration of live, attenuated vaccine within 4 weeks before the start of treatment. Note: Influenza vaccination is permitted only during influenza season, while live, attenuated influenza vaccine such as FluMist is not allowed.
* Patients receiving concurrent chemotherapy drugs,other immunosuppressive agents,or other investigational treatment.Long-term corticosteroid users are also excluded.
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Objective Response Rate | At least 6 weeks after start of treatment
  ORR was defined as the proportion of participants with partial response (PR) or complete response (CR) to treatment as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Two years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.
Objective Response Rate (ORR) in Non-irradiated Lesion | At least 6 weeks after start of treatment
  Objective Response Rate (ORR) in Non-irradiated Lesion was defined as the proportion of patients with at least 30% reduction from baseline in the longest diameter of any of non-irradiated target lesions defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at any time-point from the date of treatment initiation to the date of last follow-up.
Overall Survival | Two years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.
Progression Free Survival | Two years
  PFS was measured from the date of enrollment to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death due to any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University; Xinghao Ai, Study Director — Shanghai Chest Hospital; Zhengbo Han, Study Director — Shengjing Hospital; Qian Chu, Study Director — Tongji Hospital; Xiaorong Dong, Study Director — Union Hospital; Lin Wu, Study Director — Hunan Cancer Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Ni J, Zhou Y, Wu L, Ai X, Dong X, Chu Q, Han C, Wang X, Zhu Z. Sintilimab, stereotactic body radiotherapy and granulocyte-macrophage colony stimulating factor as second-line therapy for advanced non-small cell lung cancer: safety run-in results of a multicenter, single-arm, phase II trial. Radiat Oncol. 2021 Sep 15;16(1):177. doi: 10.1186/s13014-021-01905-3. PMID 34526044